CLINICAL TRIAL: NCT04808700
Title: Prospective Interventional Clinical Trial of an MRI Based Patient Specific Focal Knee Resurfacing Implant
Acronym: Episealer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S57685
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Focal Cartilage Lesions
Keywords: Cartilage lesions; Episealer implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focal cartilage lesion (Other): Patients with focal cartilage lesions who underwent a knee surgery using the Episealer implant
  Interventions: Other: Follow-up of Episealer implant

INTERVENTIONS:
Other: Follow-up of Episealer implant — Follow-up and radiographic evaluation in patients who received an Episealer implant

SUMMARY:
Lesions in the cartilage are common disorders. Arthroscopy lavage and debridement micro fracturing, mosaic plasticity as well as osteochondral autograft transplantation (OATS) are methods used for treatment of the lesions. Some have shown to help the patients but there is an ongoing treatment gap especially for patients with knee lesions and early osteoarthritis.

Episurf Medical has developed a Focal Knee Resurfacing (FKR) implant, the Episealer® implant. The implant is used for treatment of focal cartilage lesions of the lateral or medial femoral condyle in order to alleviate pain and improve range of motion.

In this study, the investigators aims to establish if this implant is a viable option for focal cartilage lesions of the distal femur not responding, or not eligible for, biological treatment options (eg. microfracturing)

DETAILED DESCRIPTION:
Lesions in the cartilage are common disorders. In the knee, cartilage lesions are found in over 50 % of all arthroscopies, where 25 % of these are of focal character and the majority are found in the medial femoral condyle. The quality of life of patients with focal cartilage defects is significantly affected and it has been shown that the quality of life is affected to the same extend as in patients scheduled for knee replacement. Arthroscopy lavage and debridement micro fracturing, mosaic plasticity as well as osteochondral autograft transplantation (OATS) are methods used for treatment of the lesions. Some have shown to help the patients but there is an ongoing treatment gap especially for patients with knee lesions and early osteoarthritis.

Episurf Medical has developed a Focal Knee Resurfacing (FKR) implant, the Episealer® implant. The implant is used for treatment of focal cartilage lesions of the lateral or medial femoral condyle in order to alleviate pain and improve range of motion. The implant and surgical instruments are customized to each patient's joint anatomy, position, and size of injury, based on patient-specific images (MRI).

In this study, the investigators aims to establish if this implant is a viable option for focal cartilage lesions of the distal femur not responding, or not eligible for, biological treatment options (eg. microfracturing).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a focal cartilage lesion of the distal femur in which biological surgical methods have failed or are not eligible
* Minimal age of 18 years old (Preferred age group >40 years)
* Suitable for implant, to be determined by analysis of MRI imaging. Suitability is set by the size and location of the lesion. The maximum size of the lesion is set at 6cm².
* Informed consent obtained

Exclusion Criteria:

* Active or recent (<1 yr) septic arthritis of the involved knee
* Associated symptomatic untreated ligamentary or meniscal pathology in the involved knee
* (Severe) osteoarthritis in the involved or other compartments of the involved knee
* Severe osteoporosis
* MRI not possible (eg. due to pacemaker)
* Marked valgus- or varus alignment (>6 degrees)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic and clinical evaluation | within a time frame of 2 years
  Survival of the implant up to 24 months post treatment with loss of the primary implant

CONTACTS AND LOCATIONS:
Overall Officials: Hillde Vandenneucker, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No